CLINICAL TRIAL: NCT00364130
Title: Bone Health in Pediatric Crohn's Disease: A Low Magnitude Mechanical Stimulus Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Babette Zemel, Principal Investigator, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-004906; R01DK073946 (NIH)
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Low Magnitude Mechanical Stimulus (Active Comparator): Active Low Magnitude Mechanical Stimulus
  Interventions: Device: Low magnitude mechanical stimulus
- Inactive Low Magnitude mechanical Stimulus (Placebo Comparator): Inactive, or placebo low magnitude mechanical stimulus
  Interventions: Device: Placebo (inactive) low magnitude mechanical stimulus

INTERVENTIONS:
Device: Low magnitude mechanical stimulus — 10 minute daily treatment sessions standing on the low magnitude mechanical stimulus device
  Other Names: Whole body vibration
  Arms: Active Low Magnitude Mechanical Stimulus
Device: Placebo (inactive) low magnitude mechanical stimulus — 10 minute daily treatments standing on a placebo version of a low magnitude mechanical stimulus device
  Arms: Inactive Low Magnitude mechanical Stimulus

SUMMARY:
The purpose of this 12-month double blind, placebo controlled randomized trial is to evaluate the effects of daily treatments with low magnitude mechanical stimuli on bone in 160 children with Crohn disease.

DETAILED DESCRIPTION:
Skeletal growth is characterized by increases in the size of the hard outer layer of bone (cortical bone), and the density of the inner layer of bone (trabecular or "spongy" bone). Children with Crohn disease (CD) have numerous risk factors for impaired bone accumulation, including poor growth, delayed puberty, malnutrition, glucocorticoid therapy and inflammation. We reported that children with CD had significant deficits in trabecular bone mineral density (BMD), cortical dimensions, and muscle mass; bone deficits were strongly associated with muscle deficits. No trials of therapies that build bone or prevent bone breakdown have been conducted in chronic pediatric inflammatory diseases. The capacity to increase bone mass and dimensions in response to mechanical loading is greatest during growth. Recent studies demonstrate that brief daily exposure to low magnitude mechanical stimuli (LMMS) enhances bone mass and quality. This 12-month double blind, placebo controlled randomized trial will evaluate daily 10-minute treatments with LMMS in 160 children with CD. Trabecular BMD, cortical dimensions, and muscle area will be measured by quantitative computed tomography (QCT). The LMMS device monitors adherence; these data will be transmitted by modem to the psychologist who will work closely with subjects to optimize adherence. All subjects will be provided with calcium and vitamin D supplements. The primary aims are to determine if treatment with LMMS results in increased trabecular BMD in the lower leg and spine and increased cortical dimensions in the lower leg in children with CD, compared with placebo controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-21 years
* Diagnosis of Crohn disease > 6 months
* Tibia vBMD z-score < 25th%tile for age and sex

Exclusion Criteria:

* Pregnancy
* Weight > 250 lb
* Medical illness (unrelated to Crohn)
* Cognitive/developmental disorder
* Do not speak English
* > 1 primary residence
* Unwilling to commit to 2 year study
* Sibling or cousin enrolled in trial

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2007-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babette Zemel, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began May 17, 2007 and ended June 25, 2010. Participants were recruited from the Center for Inflammatory Bowel Disease at CHOP and through referrals from physicians outside CHOP. The study was also advertised on the Crohn's and Colitis Foundation Website.
Pre-assignment Details: Patients between the ages of 8-21 years with a diagnosis of Crohn disease for at least 6 months were eligible for a screening visit. Patients meeting the entry criteria (pQCT trabecular volumetric BMD z-score below the 25th percentile)were randomly allocated 1:1 to an active LMMS device or a placebo device.
Groups:
- Active: Active Low Magnitude Mechanical Stimulus
  Low magnitude mechanical stimulus : 10 minute daily treatment sessions standing on the low magnitude mechanical stimulus device
- Pacebo: Placebo (inactive) low magnitude mechanical stimulus : 10 minute daily treatments standing on a placebo version of a low magnitude mechanical stimulus device
Period: Intervention Period
Arm/Group | Active | Pacebo
Started | 69 | 69
Completed | 60 | 61
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 4 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5
Period: Post Intervention Follow-up Period
Arm/Group | Active | Pacebo
Started | 60 | 61
Completed | 55 | 50
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Pacebo | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 63 | 63 | 126
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.11475 (2.900821) | 14.51452 (2.720447) | 14.3134 (2.816848)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 36 | 36 | 72
Region of Enrollment [Number; unit: participants]
  United States | 69 | 69 | 138

OUTCOME MEASURES:

1. Primary Outcome: Change in Tibia Trabecular Volumetric Bone Mineral Density (BMD) Z-score at 12 Months
Description: We calculated the mean change in tibia trabecular volumetric BMD Z-score between baseline and 12 months, as measured by peripheral quantitative computed tomography (pQCT).
  The Z-score, or Standard Deviation Score, is a measure of the number of standard deviations that an individual is above or below the median value in a healthy child or adolescent of the same age, sex and race. For example, a Z-score of 0 means that an individual's result is equivalent to the 50th percentile in a healthy population. A Z-score of -1.0 means that an individual's result is equovalent to the 16th percentile in a healthy population.
Time Frame: 12 months
Population: The number was determined by the number of participants with measures at both baseline and 12 month time points. The analysis was intention to treat.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active | Pacebo
Number analyzed (Participants) | 60 | 61
Z-score | 0.15 (0.55) | 0.23 (0.70)
Statistical Analysis 1: Comparison: Active vs Pacebo; Test type: Superiority or Other; p = 0.38, Regression, Linear — The outcome is not adjusted for multiple comparisons

2. Primary Outcome: Change in Tibia Cortical Area Z-score 12 Months
Description: We calculated the mean change in tibia cortical area Z-score, as measured by pQCT, between baseline and 12 months.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active | Pacebo
Number analyzed (Participants) | 60 | 61
Z-score | 0.17 (0.58) | 0.20 (0.59)
Statistical Analysis 1: Comparison: Active vs Pacebo; Test type: Superiority or Other; p = 0.80, Regression, Linear — The outcome is not adjusted for multiple comparisons

3. Primary Outcome: Change in Spine Volumetric BMD Z-score at 12 Months
Description: We calculated the mean change in spine volumetric BMD Z-score, as measured by QCT, between baseline and 12 months
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active | Pacebo
Number analyzed (Participants) | 60 | 61
Z-score | 0.22 (0.59) | -0.02 (0.67)
Statistical Analysis 1: Comparison: Active vs Pacebo; Test type: Superiority or Other; p = 0.02, Regression, Linear — The outcome is not adjusted for multiple comparisons

4. Secondary Outcome: Change in Posteroanterior Lumbar Spine Areal BMD Z-score
Description: We calculated the mean change in posterior anterior lumbar spine areal BMD Z-score between baseline and 12 months as measured by DXA
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active Low Magnitude Mechanical Stimulus | Inactive Low Magnitude Mechanical Stimulus
Number analyzed (Participants) | 60 | 61
Z-score | 0.20 (0.44) | 0.09 (0.44)
Statistical Analysis 1: Comparison: Active Low Magnitude Mechanical Stimulus vs Inactive Low Magnitude Mechanical Stimulus; Test type: Superiority or Other; p = 0.27, Regression, Linear — The outcome was not adjusted for multiple comparisons

5. Secondary Outcome: Change in Total Hip Areal BMD Z-score Between Baseline and 12 Months
Description: We calculated the mean change in total hip bone mineral density z-score, as measured by DXA, between baseline and 12 months
Time Frame: 12months
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active | Pacebo
Number analyzed (Participants) | 60 | 61
Z-score | 0.24 (0.44) | 0.25 (0.43)
Statistical Analysis 1: Comparison: Active vs Pacebo; Test type: Superiority or Other; p = 0.84, Regression, Linear — The outcome is not adjusted for multiple comparisons

6. Secondary Outcome: Change in Femoral Neck Areal BMD Z-score Between Baseline and 12 Months
Description: We calculated the mean change in femoral neck areal bmd Z-score between baseline and 12 months as measured by DXA
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active | Pacebo
Number analyzed (Participants) | 60 | 61
Z-score | 0.19 (0.45) | 0.22 (0.45)
Statistical Analysis 1: Comparison: Active vs Pacebo; Test type: Superiority or Other; p = 0.66, Regression, Linear — The outcome is not adjusted for multiple comparisons

7. Secondary Outcome: Change in Whole Body Bone Mineral Content Z-score Between Baseline and 12 Months
Description: We calculated the mean change in whole body bone mineral content Z-score, as measured by DXA, between baseline and 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Active | Pacebo
Number analyzed (Participants) | 60 | 61
Z-score | 0.20 (0.40) | 0.18 (0.43)
Statistical Analysis 1: Comparison: Active vs Pacebo; Test type: Superiority or Other; p = 0.70, Regression, Linear — The outcome is not adjusted for multiple comparisons

8. Secondary Outcome: Change in QCT Tibia Trabecular Volumetric BMD at 12 Months
Description: We calculated the mean change in tibia trabecular volumetric BMDbetween baseline and 12 months as measured by (QCT)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Active | Pacebo
Number analyzed (Participants) | 60 | 61
cm^3 | 1.05 (10.5) | 1.35 (12.93)
Statistical Analysis 1: Comparison: Active vs Pacebo; Test type: Superiority or Other; p = 0.98, Regression, Linear — Outcome is not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 6 months, 1 year and 2 years.
Arm/Group | Active | Pacebo
Serious Adverse Events (participants affected / at risk) | 7/69 | 6/69
Other Adverse Events (participants affected / at risk) | 10/69 | 10/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=69) | Pacebo (N=69)
hospitalization for infection (Infections and infestations) | 5 (6) | 5 (5) — hospitalization for various infectsion: pneumonia, viral infection, cellulitis, clostridium difficile infection.
hospitalization for for appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization for migraine headache (Nervous system disorders) | 1 (4) | 0 (0)
hospitalization for small bowel overgrowth (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=69) | Pacebo (N=69)
headache (Nervous system disorders) | 1 (1) | 4 (4)
abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
stool changes (Gastrointestinal disorders) | 5 (5) | 1 (1) — increased frequency, urgency, increased loose stools/diarrhea
lower extremity pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) — knee, leg, ankle or foot pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No